CLINICAL TRIAL: NCT03112356
Title: The Value of 99mTc-Leukoscan® Scintigraphy in the Diagnosis of Infectious Endocarditis on Surgical Materials
Acronym: PLEIM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0728
Record Dates: First submitted 2017-03-24; First posted 2017-04-13 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Endocarditis
Keywords: infectious endocarditis; prosthetic valve infection; implantable cardiac device infection; 99mTc-Leukoscan® scintigraphy
MeSH Terms: conditions — Endocarditis; Endocarditis, Subacute Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-Leukoscan® scintigraphy (Experimental): Patients presenting a suspicions of infectious endocarditis on surgical materials and undergoing the 99mTc-Leukoscan® scintigraphy
  Interventions: Drug: 99mTc-Leukoscan® scintigraphy

INTERVENTIONS:
Drug: 99mTc-Leukoscan® scintigraphy — Gated single photon emission computed tomography with co-registered computer tomography (gated SPECT-CT) 6 hours and 24 hours after infusion of 99mTc-Leukoscan (1000 MBq)

SUMMARY:
Infectious endocarditis is a serious pathology with difficult diagnosis especially on prosthetic valves or cardiac device because of the plurality of clinical presentations and the low sensitivity value of echocardiography in these patients. Despite a well validated indication for the detection of septic emboli, the value of FDG-PET for the detection of prosthetic valves or cardiac implantable device is still unclear especially because of frequent non-septic inflammatory processes.

To improve the specificity value, the use of radio-labeled leukocytes scintigraphy is conventionally proposed. An alternative method is to label leukocytes in vivo with an anti-murin anti body fragment ( Sulesomab , Leukoscan®). This scintigraphy is regularly used in the investigation of osteomyelitis and has been proposed in infectious endocarditis. To knowledge of investigators, the value of Leukoscan® scintigraphy on prosthetic valve or cardiac device infection had not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged > 21 years
* Patients presenting a suspicions of infectious endocarditis on surgical materials
* Written informed consent

Exclusion Criteria:

* Patient with a history of exposure to murine antigens, particularly a patient who has already received a 99mTc-Leukoscan® scintigraphy
* Patients whose clinical condition requires prompt care, not allowing them to wait for the examination
* Pregnant or nursing (including pumping for storage and feeding)
* Patients under adapted antibiotic therapy for more than 15 days
* Deprivation of civil rights (curatorship, guardianship, safeguard of justice)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-10-14 (Estimated); Study Completion 2018-10-14 (Estimated)

PRIMARY OUTCOMES:
Presence or not of infectious endocarditis on surgical materials | 3 months (plus or minus 1 month)
  The presence or not of infectious endocarditis on surgical materials will be measured using Duke's criteria of patients follow-up at 3 months (plus or minus 1 month).

CONTACTS AND LOCATIONS:
Overall Officials: Bastien GREGOIRE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No